CLINICAL TRIAL: NCT01727375
Title: Prevention of Delirium With Light in the Intensive Care Unit
Acronym: PreDeLight-ICU
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Univ.-Prof. Dr. Claudia Spies, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PreDeLight-ICU
Record Dates: First submitted 2012-07-04; First posted 2012-11-16 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Delirium
Keywords: delirium, light, ICU, sleep
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard light (No Intervention): In this arm patients receive standard lightening conditions
- Ciradian light (Experimental): In this arm patients receive artificial ceiling light (circadian light) at the bedside.
  Interventions: Other: Circadian light

INTERVENTIONS:
Other: Circadian light — Artificial ceiling lighting throughout the day will be provided by the Philips HealWell system, CE marked, which is able to deliver varying light levels and warmer or cooler light according to the time of the day (circadian light). Emergency or examination lighting can be set on demand as circumstances require.
  Lighting conditions at the patients bedside will be characterized by transformations on the time-series of light levels as measured by a luxmeter. The following metrics will be used for lighting characterization in a period of 24h: mean levels of bright and dark periods, contrast between bright and dark periods, clustering of bright and dark periods, and circadian variation.
  Arms: Ciradian light

SUMMARY:
The purpose of this multicenter randomised controlled trial is to investigate if circadian light at the patients bedside (using Philips HealWell system, CE marked)significantly reduces prevalence of delirium in mechanically ventilated intensive care unit patients.

DETAILED DESCRIPTION:
Patients, who are randomly assigned to the "Lightening arm" will have the circadian light for the whole ICU stay. Light levels at the patients bedside will be measured continuously: embedded light sensors provide irradiance and luminous lux recordings in red, green, and blue color bands and a white light measurement in lux

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with age 18 years and above
* Intensive Care Unit stay ≥ 48 hours
* Invasive mechanical ventilation or not invasive mechanical ventilation (with positive ventilation pressure >6hours/day and highflow >30 litres) on the day of Intensive Care Unit admission

Exclusion Criteria:

* Patients with a history Intensive Care Unit stay during the actual hospital stay
* Patients with delirium on the day of Intensive Care Unit admission
* Patients with psychiatric diseases
* Patients with a history of stroke and known cognitive dysfunctions
* Participation in other clinical studies 10 days before study inclusion and during the study period
* Psychiatric disease
* History of stroke with known residual cognitive deficits
* History of Asystolia or pulseless electric activity with cardiopulmonary resuscitation during entire hospital stay
* Analphabetism
* Unability of German language use
* Anacusis or Hypoacusis with hearing aid device, Amaurosis
* Allergies to any ingredient of the electrode fixing material
* Lacking willingness to save and hand out data within the study
* Accommodation in an institution due to an official or judicial order
* The informed consent of the patient or the subject's legally acceptable representative can´t be obtained in time
* Patient has a power of attorney or patient's provision, where he/she refuses participation in any clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Prevalence of delirium | Participants will be followed for the duration of Intensive Care Unit stay, an expected average of 5 days
  Dekirium will be measured with the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU)

SECONDARY OUTCOMES:
Delirium prevalence | Participants will be followed for the duration of Intensive Care Unit stay, an expected average of 5 days
  In this case, delirium will be measured with the help of the Intensive care Delirium Screening Checklist (ICDSC)
Severity of delirium | Participants will be followed for the duration of Intensive Care Unit stay, an expected average of 5 days
  Severity of delirium will be measured with the help of the Intensive Care Delirium Screening Checklist (ICDSC)
Duration of delirium | Participants will be followed for the duration of Intensive Care Unit stay, an expected average of 5 days
Prevalence of subsyndromal delirium (SSD) | Participants will be followed for the duration of Intensive Care Unit stay, an expected average of 5 days
Severity of anxiety | Participants will be followed for the duration of Intensive Care Unit stay, an expected average of 5 days
Cognitive Dysfunction | ICU admission, ICU discharge, 6 months after hospital discharge, 12 months after ICU discharge
Post-Traumatic Stress Disorder (PTSD) | 6 and 12 months after hospital discharge
Sleep quality | In the night, starting 48 hours after ICU admission
ICU length of stay | Participants will be followed for the duration of Intensive Care Unit stay, an expected average of 5 days
Duration of mechanical ventilation | Participants will be followed for the duration of Intensive Care Unit stay, an expected average of 5 days
Hospital length of stay | Participants will be followed for the duration of Intensive Care Unit stay, an expected average of 4 weeks
Level of sedation | Participants will be followed for the duration of Intensive Care Unit stay, an expected average of 5 days
Pain level | Participants will be followed for the duration of Intensive Care Unit stay, an expected average of 5 days
Amount of administered opioids | Participants will be followed for the duration of Intensive Care Unit stay, an expected average of 5 days
Amount of administered benzodiazepines | Participants will be followed for the duration of Intensive Care Unit stay, an expected average of 5 days
Amount of administered sedatives | Participants will be followed for the duration of Intensive Care Unit stay, an expected average of 5 days
Amount of administered antipsychotics | Participants will be followed for the duration of Intensive Care Unit stay, an expected average of 5 days
Mortality | ICU discharge, hospital discharge, 6 months after hospital discharge, 12 months after hospital discharge
Light levels (lux) Light levels (lux) | Participants will be followed for the duration of Intensive Care Unit stay, an expected average of 5 days
Light frequencies | Participants will be followed for the duration of Intensive Care Unit stay, an expected average of 5 days
Noise levels (decibel) | Participants will be followed for the duration of Intensive Care Unit stay, an expected average of 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Dept. of Anesthesiology and Intensive Care Medicine, CVK/CCM, Charité - Universitaetsmedizin Berlin
Locations (1):
- Center of Sleep Medicine, Campus Charité Mitte, Charité - Universitaetsmedizin, Berlin, State of Berlin, Germany